CLINICAL TRIAL: NCT01021163
Title: Effects of N-acetylcysteine on Pulmonary Function in High-risk Patients Undergoing Off-pump Coronary Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Young Lan Kwak / Professor, Anesthesiology and Pain Medicine
Model: Parallel | Purpose: Treatment
Other Study IDs: 4-2007-0236
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Artery Occlusion
MeSH Terms: conditions — Coronary Occlusion | interventions — Acetylcysteine; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-acetylcysteine , saline (Placebo Comparator)
  Interventions: Drug: N-acetylcysteine, saline

INTERVENTIONS:
Drug: N-acetylcysteine, saline — Inject 100 mg/kg of N-acetylcysteine or the equivalent amount of saline for 15 minutes before the skin incision, then continuously inject 40 mg/kg/day of N-acetylcysteine or the equivalent amount of saline during the next 24 hours.

SUMMARY:
The purpose of this study is to study the effects of N-acetylcysteine on pulmonary function in high-risk patients undergoing off-pump coronary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Euroscore ≥ 5

Exclusion Criteria:

* Patients in need of emergency surgery,acute renal failure patients, kidney transplanted patients, patients injected with NAC 5days before planned surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea